CLINICAL TRIAL: NCT06906822
Title: A Phase II, Open-label, Multicenter, Non-Randomized Study of the Efficacy and Safety of Enfortumab Vetodin in Combination With Pembrolizumab Previously Treated Advanced Melanoma
Brief Title: PLUG-IN: Pembrolizumab Combined With Enfortumab Vedotin for Advanced Melanoma Patients
Acronym: PlugIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM 2303; 2024-514163-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: Melanoma; Enfortumab; vedotin; pembrolizumab
MeSH Terms: conditions — Melanoma | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, non-randomized open-label, 2-cohort, phase 2 study to evaluate the ORR of pembrolizumab in combination with enfortumab vedotin (EV) in previously treated participants with unresectable stage III or IV melanoma and disease progression on standard therapy.
  A total of 60 patients will be enrolled after signing the informed consent in two different cohorts:
  Cohort 1: patients who did not have BRAF mutation V600E and had disease progression on immune (IO) therapy.
  Cohort 2: patients with activating BRAF mutations, must have progressed on IO therapy and BRAF/MEKi
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): patients who did not have BRAF mutation V600E and had disease progression on immune (IO) therapy.
  Interventions: Drug: enfortumab vedotin; Drug: pembrolizumab
- Cohort 2 (Experimental): patients with activating BRAF mutations, must have progressed on IO therapy and BRAF/MEKi
  Interventions: Drug: enfortumab vedotin; Drug: pembrolizumab

INTERVENTIONS:
Drug: enfortumab vedotin — Enfortumab vedotin 1.25 mg/kg be administered on Days 1,8,22 and 29 of every 6-week cycle by IV infusion given over approximately 30 minutes.
Drug: pembrolizumab — Pembrolizumab 400 mg on day 1 of each 42-day cycle (Q6W)

SUMMARY:
There is a lack of strategies for patients who progress after responding to PD-1/l-1 in melanoma. High expression of Nectin4 in skin and melanomas may serve as a new target in advanced melanomas. The combination of enfortumab/vedotin (EV) and pembrolizumab has shown synergistic effect in various solid tumors. Enfortumab vedotin and pembrolizumab may have a dual effect on clinical outcomes.

PLUGIN is a multicenter, non-randomized open-label, 2-cohort, phase 2 study to evaluate the ORR of pembrolizumab in combination with enfortumab vedotin (EV) in previously treated participants with unresectable stage III or IV melanoma and disease progression on standard therapy.

The primary objective is evaluate the efficacy of enfortumab/vedotin and pembrolizumabplus pembrolizumab in advanced melanoma.

Hypothesis: 1) High expression of Nectin4 in skin and melanomas may serve as a new target in advanced melanomas; 2)EV+Pembrolizumab has shown synergistic effect in various solid tumors; 3) There is a lack of strategies for patients who respond to PD1-mAbs in melanoma.

Primary Endpoint: Objective Response Rate (ORR) as assessed by the investigator according RECIST 1.1

A total of 60 patients will be enrolled in this study to evaluate efficacy and outcomes in two different cohorts:

Cohort 1: patients who did not have BRAF mutation V600E and had disease progression on immune (IO) therapy.

Cohort 2, patients with activating BRAF mutations, must have progressed on IO therapy and BRAF/MEKi

DETAILED DESCRIPTION:
1. RATIONALE

   There is a lack of strategies for patients who progress after responding to PD-1/l-1 in melanoma. High expression of Nectin4 in skin and melanomas may serve as a new target in advanced melanomas. The combination of enfortumab vedotin and pembrolizumab has shown synergistic effect in various solid tumors. Enfortumab vedotin and pembrolizumab may have a dual effect on clinical outcomes:
   1. Enfortumab vedotin could induce a tumor response based on a high dose of the microtubule disruptor in tumor cells.
   2. Enfortumab vedotin could enhance antitumor immunity and prolong the benefit of continuous PD1 therapy.
2. OBJECTIVE(S), HYPOTHESIS(ES), AND ENDPOINT(S)

2.1 Primary Objective(s), Hypothesis(es), and Endpoint(s) Objective: This study will evaluate the efficacy of EV plus pembrolizumab in advanced melanoma.

Hypothesis: 1) High expression of Nectin4 in skin and melanomas may serve as a new target in advanced melanomas; 2)EV+Pembrolizumab has shown synergistic effect in various solid tumors; 3) There is a lack of strategies for patients who respond to PD1-mAbs in melanoma.

The combination of EV+Pembrolizumab may have a dual effect on outcomes:

1. EV could induce a tumor response based on a high dose of the microtubule disruptor in tumor cells.
2. EV could enhance antitumor immunity and prolong the benefit of continuous PD1 therapy.

   Primary Endpoint:

   - Objective Response Rate (ORR) as assessed by the investigator through Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study.

   2.2 Secondary Objective(s), Hypothesis(es), and Endpoint(s)

   Secondary Endpoint:

   - Progression-free Survival (PFS) as assessed by RECIST 1.1. PFS is defined as the time from first dose of study treatment to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first.
   * Overall Survival (OS), defined as the time from first dose of study treatment to the date of death from any cause.
   * Clinical Benefit Rate (CBR), defined as proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST V1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a CBR event.
   * Duration of Response (DoR) as Assessed by RECIST 1.1. DoR is considered an acceptable measure of clinical benefit when considered with ORR.
   * Treatment-free Survival (TFS), defined as the time from the end of study treatment until the start of subsequent treatment, progression or death, whichever occurs first.
   * Treatment-free Interval (TFI), defined as the time from the end study treatment until the start of subsequent treatment.
   * The safety objective for this study is to evaluate the safety of EV plus pembrolizumab on the basis of the following endpoints:

     1. Number of Participants with Adverse Events (AEs) Safety Objective Incidence and severity of adverse events, with severity determined according to b. National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

     c. Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs)
   * Mean change from baseline in health-related quality of life (HRQoL) scores as assessed through use of the two-item global health status (GHS)/HRQoL subscale of the European Organisation for Research and Treatment of Cancer Quality ofLifeCore 30 (EORTC QLQ-C30) at specified time points.

   2.3. Exploratory Objective(s) Objective: Correlative studies (microbiome and transcriptomic analysis)

   5. TRIAL DESIGN This is a multicenter, non-randomized open-label, 2-cohort, phase 2 study to evaluate the ORR of pembrolizumab in combination with enfortumab vedotin (EV) in previously treated participants with unresectable stage III or IV melanoma and disease progression on standard therapy.

   Specific procedures to be performed during the study, as well as their prescribed times and associated visit windows, are specifically outlined in the protcolo.

   The study will include a Screening Phase, a Treatment Phase, and a Posttreatment Follow-Up Phase. The Screening Phase assessments must be performed within 30 days before randomization. Potential participants will be screened to determine if they meet the required eligibility criteria.

   Assessments will include AE monitoring, concomitant medication review, physical examination and ophthalmological examination, vital signs, blood pressure, ECG, hematology, chemistry, urine dipstick, and ECOG performance status.

   6. TRIAL POPULATION

   A total of 60 patients will be enrolled after signing the informed consent in two different cohorts:

   - Cohort 1: patients who did not have BRAF mutation V600E and had disease progression on immune (IO) therapy.

   - Cohort 2: patients with activating BRAF mutations, must have progressed on IO therapy and BRAF/MEKi.

   Patients are males/females, ≥18 years old, with measurable disease according to RECIST 1.1 and progressive disease / recurrence documented within 12 weeks from the last dose of previous anti-PD-1/L1. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, have recovered from previous toxicities and with an adequate organ function. Archival tumor tissue sample or newly obtained biopsy is requested. Patients with contraindications to receive immunotherapy, exposed previously to enfortumab vedotin and pregnant or breastfeeding women are excluded.

   7. STUDY TREATMENTS

   Enfortumab vedotin will be administered on Days 1, 8, 22 and 29 of every 6-week cycle by IV infusion given over approximately 30 minutes. Pembrolizumab 400 mg will be administered as a 30 minute IV infusion every 6 weeks.

   Enfortumab vedotin will be administered until progression of the disease, lack of benefit, death, consent withdrawal or unacceptable toxicity. Treatment with pembrolizumab will last a maximum of 18 cycles. Pembrolizumab may be discontinued earlier in case of progression of the disease, lack of benefit, death, consent withdrawal or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of unresectable or metastatic melanoma will be enrolled in this study.
2. Participants must have measurable disease by investigator assessment according to RECIST v1.1 Participants with prior definitive radiation therapy must have measurable disease per RECIST v1.1 that is outside the radiation field or has demonstrated unequivocal progression since completion of radiation therapy.
3. Male participants:

   a. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for 9 months after last dose of EV or 4 months after pembrolizumab, whichever occurs last; and refrain from donating sperm during this period.
4. Female participants:

   A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3. OR
   2. WOCBP should remain on contraception for 12 months after the last dose of EV or 4 months after pembrolizumab, whichever occurs last.
5. Participants must have received prior systemic therapy for locally advanced or metastatic melanoma:

   a. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria: i. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   * Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1.
   * The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression.

   ii. Progressive disease / recurrence has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb. Progressive disease is determined according to iRECIST. This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.

   b. BRAF mutated patients should have received BRAF/MEK inhibitors and PD1/PDL1 therapy c. Prior CTLA4 therapy is allowed.
6. Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.

   Note: Patients who had cutaneous adverse events grade 3 or superior are not eligible for the study.
7. Provide representative formalin-fixed paraffin-embedded/FFPE paraffin block obtained after last treatment progression. Patients who have no archival tumor tissue after the last treatment progression will be required to provide a fresh biopsy, if the procedure is feasible and safe for the patient. Older archival tumor samples are allowed for patients with no recent archival tissue (after last treatment progression) and not capable of undergoing a new tumor biopsy before the first dose of study treatment.. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
9. Have adequate organ function as defined in the following table (see Table 3 in protocol). Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. Participants are excluded from the study if any of the following criteria apply:

   A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Participants who have previously received enfortumab vedotin or other MMAE-based ADCs.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the scheduled date of starting the study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.

   Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease, with a 1-week washout, is permitted.
5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
6. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
7. Participants with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms that are not otherwise explained.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Known additional malignancy that is progressing or has required active treatment within the past 2 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
10. Has known active CNS metastases and/or carcinomatous meningitis. Note: Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
11. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients. Participants with known severe (≥ Grade 3) hypersensitivity to any enfortumab vedotin excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20).
12. Participants with active keratitis or corneal ulcerations. Participants with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
14. Participants with conditions requiring systemic doses of corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded.
15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required corticosteroids or has current pneumonitis/interstitial lung disease.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV) infection.
18. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:

    Known history of HBV and HCV infection As mandated by local health authority
19. Has not adequately recovered from major surgery or has ongoing surgical complications.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of contraception period.
23. Has had an allogenic tissue/solid organ transplant.
24. History of Clinical Tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period,period, from initiation of treatment up to 2 years
  Objective Response Rate (ORR) as assessed by the investigator through Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study.
  Estimates of the ORR along with the associated 95% exact binomial confidence intervals will be provided. The binomial probability that the observed melanoma ORR is > 0.15 will be calculated. Best confirmed response will be summarized. Response of melanoma will be measured by CT or MRI and assessed according to RECIST 1.1 by the investigator. If there are no assessments, the response will be taken to be unconfirmed and a non-response. Changes in tumor size from baseline will be calculated and displayed graphically, where appropriate.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) 6 months | Throughout the study period, from initiation of treatment up to 6 months
  Progression-free Survival (PFS) defined as the time from the start of treatment to disease progression or death from any cause, whichever occurs first. The PFS will be estimated by the Kaplan-Meier method. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without event will be censored on the date of first dose of the subsequent anticancer treatment. PFS will be displayed graphically where appropriate.
  PFS will be assessed by the median / mean (95% CI) and for different timepoints:
  Proportion of patients without progression at the end of follow-up. Proportion of patients at 6-months, 12-months and as deemed opportune by the time of the analysis.
  Confidence intervals (CIs) for the 25th, 50th and 75th percentiles will be reported. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable.
Progression-free Survival (PFS) 12 months | Throughout the study period, from initiation of treatment up to 12 months
  Progression-free Survival (PFS) defined as the time from the start of treatment to disease progression or death from any cause, whichever occurs first. The PFS will be estimated by the Kaplan-Meier method. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without event will be censored on the date of first dose of the subsequent anticancer treatment. PFS will be displayed graphically where appropriate. PFS will be assessed by the median / mean (95% CI) and for different timepoints: Proportion of patients without progression at the end of follow-up. Proportion of patients at 6-months, 12-months and as deemed opportune by the time of the analysis.
  Confidence intervals (CIs) for the 25th, 50th and 75th percentiles will be reported. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable.
Overall survival (OS) | Throughout the study period, from initiation of treatment up to 12 months
  Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact. OS will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. Confidence intervals (CIs) for the 25th, 50th and 75th percentiles will be reported. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable. OS will be calculated as median / mean (95% CI) and OS rate for different timepoints deemed appropriate at the time of the analysis (i.e.1-year OS rate) will also be calculated.
Overall survival (OS) | Throughout the study period, from initiation of treatment up to 24 months
  Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact. OS will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. Confidence intervals (CIs) for the 25th, 50th and 75th percentiles will be reported. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable. OS will be calculated as median / mean (95% CI) and OS rate for different timepoints deemed appropriate at the time of the analysis (i.e.1-year OS rate) will also be calculated.
Clinical Benefit Rate (CBR) | Throughout the study period, from initiation of treatment up to 24 months
  Clinical Benefit Rate (CBR): Assessed locally by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1. CBR will include the percentage/proportion of patients with CR, PR, or SD (maintained > 4 months) as their overall best response throughout the study period. The CBR will be estimated by binomial proportion, dividing the number of patients with CR, PR or SD for at least 4 months for CBR by the total number of patients studied in the population. The corresponding exact 2-sided 95% CIs will be provided. Changes in tumor size from baseline will be calculated and displayed graphically, where appropriate.
Duration of Response (DoR): | Throughout the study period, from initiation of treatment up to 12 months
  Duration of Response (DoR): The DoR will be calculated for patients who achieve a CR or PR. Dates of progression and censoring for DoR will be determined as described for PFS. Kaplan-Meier methods will be used to estimate the distribution of DoR. Quartiles including the median will be estimated by KM method along with their 95% confidence intervals.
Treatment-free Survival (TFS) | Throughout the study period, from initiation of treatment up to 24 months
  Treatment-free Survival (TFS): defined as the time from the end of study treatment until the start of subsequent treatment, progression or death, whichever occurs first, will be determined as described for PFS. Kaplan-Meier methods will be used to estimate TFS.
Treatment-free Interval (TFI) | Throughout the study period, from initiation of treatment up to 24 months
  Treatment-free Interval (TFI): defined as the time from the end of study treatment until the start of subsequent treatment; will be determined as described for PFS. Kaplan-Meier methods will be used to estimate TFI.
Adverse Events (AEs) Safety Objective | Throughout the study period, from the inclusion of the first patient up to 24 months
  Number of Participants with Adverse Events (AEs)
Incidence and severity of adverse events | Throughout the study period, from the inclusion of the first patient up to 24 months
  Incidence and severity of adverse events, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Discontinue Study Treatment Due to Adverse Events (AEs) | Throughout the study period, from the inclusion of the first patient up to 24 months
  Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo de Velasco, M.D., Ph.D., Study Director — Hospital Universitario 12 de Octubre; Ainara Soria, M.D., Ph.D., Study Director — Hospital Universitario Ramón y Cajal
Locations (13):
- Spain (13):
  - Complexo Hospitalario Universitario de A Coruña, A Coruña, A Coruña
  - Institut Català D'Oncologia - Badalona, Badalona, Barcelona
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No